CLINICAL TRIAL: NCT04113616
Title: An Open-Label, Multicenter, Phase 1b/2 Study of the Safety and Efficacy of KRT-232 When Administered Alone and in Combination With Low-Dose Cytarabine (LDAC) or Decitabine in Patients With Acute Myeloid Leukemia (AML)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: In September 2023, the study was terminated because of a Sponsor decision, unrelated to safety concerns.
Sponsor: Kartos Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KRT-232-104
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Relapsed or Refractory Acute Myeloid Leukemia (AML); Acute Myeloid Leukemia (AML), Secondary to Myeloproliferative Neoplasms (MPN)
Keywords: navtemadlin
MeSH Terms: conditions — Recurrence; Leukemia, Myeloid, Acute | interventions — navtemadlin; 2-((3R,5R,6S)-5-(3-chlorophenyl)-6-(4-chlorophenyl)-1-((S)-1-(isopropylsulfonyl)-3-methylbutan-2-yl)-3-methyl-2-oxopiperidin-3-yl)acetic acid; Cytarabine; Decitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A - Arm 1 (Experimental): KRT-232+LDAC:
  KRT-232 will be administered orally, once daily (QD), on Days 1-7 in combination with LDAC administered at 20 mg/m2/day subcutaneously on Days 1-10 in a 28-day cycle.
  Interventions: Drug: KRT-232; Drug: Cytarabine
- Part A - Arm 2 (Experimental): KRT-232(7-Day)+Decitabine:
  KRT-232 will be administered orally, once daily (QD), on Days 1-7 in combination with Decitabine administered at 20 mg/m2/day intravenously on Days 1-5 in a 28-day cycle.
  Interventions: Drug: KRT-232; Drug: Decitabine
- Part A - Arm 3 (Experimental): KRT-232(14-Day)+Decitabine:
  KRT-232 will be administered orally, once daily (QD), on Days 1-7 and Days 15-21 (7 days on/7 days off/7 days on/7 days off) in combination with Decitabine administered at 20 mg/m2/day intravenously on Days 1-5 in a 28-day cycle.
  Interventions: Drug: KRT-232; Drug: Decitabine
- Part B - Arm 1 (Experimental): KRT-232 administered at 360 mg orally, once daily (QD) on Days 1-7 with 21 days off on a 28-day treatment cycle
  Interventions: Drug: KRT-232
- Part B - Arm 2 (Experimental): KRT-232 administered at 360 mg orally, once daily (QD) on Days 1-7 with 21 days off on a 28-day treatment cycle in Cycle 1, followed by 240 mg orally, once daily (QD) on Days 1-7 with 21 days off on a 28-day cycle, in the subsequent cycles.
  Interventions: Drug: KRT-232
- Part B - Arm 3 (Experimental): KRT-232 administered at 180 mg orally, once daily (QD) on Days 1-7 with 14 days off on a 21-day treatment cycle.
  Interventions: Drug: KRT-232

INTERVENTIONS:
Drug: KRT-232 — KRT-232 is an experimental MDM2 inhibitor anti-cancer drug taken by mouth.
Drug: Cytarabine — Cytarabine is an anti-cancer chemotherapy drug taken via injection.
  Other Names: cytosine arabinoside; Cytosar-U; Depocyt; Arabinosylcytosine; Ara-C
  Arms: Part A - Arm 1
Drug: Decitabine — Decitabine is an anti-cancer chemotherapy drug taken via injection.
  Other Names: Dacogen
  Arms: Part A - Arm 2; Part A - Arm 3

SUMMARY:
This study evaluates KRT-232, a novel oral small molecule inhibitor of MDM2, when administered alone and in combination with low-dose cytarabine (LDAC) or Decitabine for the treatment of adults with Acute Myeloid Leukemia (AML) and AML secondary to myeloproliferative neoplasms (MPN). Participants must be relapsed/refractory (having failed prior therapy) and will be assigned to receive monotherapy (KRT-232 alone) or combination therapy (KRT-232 with LDAC or KRT-232 with Decitabine).

ELIGIBILITY:
Key Inclusion Criteria:

* Part A: Patients with relapsed or refractory AML, or newly-diagnosed AML secondary to MPN
* Part B:Patients with relapsed or refractory AML secondary to MPN (myelofibrosis [MF], polycythemia vera [PV], or essential thrombocythemia [ET]); patients may have been treated with ≥1 prior lines of therapy for their AML secondary to MPN.
* Adequate hepatic and renal function
* Appropriate prior treatment with an FLT3 or IDH1/2 inhibitor where applicable

Key Exclusion Criteria:

* Patients who are TP53 mutation positive
* Prior treatment with an MDM2 antagonist therapy
* Patients treated with ≥ 18 g/m2 of cytarabine within the prior 90 days are not eligible to be treated with cytarabine on this study but may be treated with decitabine (for Part A) .
* Patients previously treated with decitabine are not eligible to receive decitabine on this study but may be treated with cytarabine (for Part A) .
* Patients who have received an allogeneic HSCT within 90 days of enrollment or who have active graft-versus-host disease requiring active therapy (for Part A)
* Allogeneic stem cell transplant within 3 months; autologous stem cell transplant within 3 months or active graft-versus-host disease prior to first dose of study treatment (for Part B)
* Patients who have received immunosuppressive therapy for graft-versus-host disease within 1 month prior to enrollment into this study
* Patients who are eligible for an allogeneic HSCT per the opinion of the investigator and have a donor. Patients who are HSCT-eligible in the opinion of the investigator, but who refuse a transplant, are eligible for the study.
* Patients with known CNS involvement with AML, acute promyelocytic leukemia (APL), or a history of bleeding diathesis
* Patients who have had major surgery within 28 days prior to the first treatment with KRT-232
* Women who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
Part A: To determine KRT-232 recommended phase 2 dose (RP2D) | 28 Days
  Number of dose-limiting toxicities (DLTs) of KRT-232 in combination with cytarabine or decitabine
Part B: To determine the RP2D of KRT-232 | 2 years after last patient enrolled
  The safety review committee (SRC) will determine the RP2D based on safety and tolerability data obtained from each arm

SECONDARY OUTCOMES:
Part A: To determine the rates of complete remission (CR) and complete remission with partial hematological improvement (CRh) | 12 weeks
  Proportion of patients achieving complete remission (CR) or complete remission with partial hematological improvement (CRh) as determined by Modified 2017 European LeukemiaNet (ELN) response criteria
Part B: To determine the rates of complete remission (CR), CR with partial hematological improvement (CRh) and CR with incomplete hematologic recovery (CRi) | 12 weeks
  Proportion of patients achieving complete remission (CR), complete remission with partial hematological improvement (CRh), and CR with incomplete hematologic recovery (CRi) as determined by Modified 2017 European LeukemiaNet (ELN) response criteria

CONTACTS AND LOCATIONS:
Locations (59):
- United States (8):
  - University of Chicago, Chicago, Illinois
  - University of Maryland Medical Center, Baltimore, Maryland
  - Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Weill Cornell, New York, New York
  - The Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
- Australia (5):
  - Monash Health, Clayton
  - St. George Hospital, Kogarah
  - Royal Perth Hospital, Perth
  - Calvary Mater Newcastle Hospital, Waratah
  - Perth Blood Institute, West Perth
- Belgium (5):
  - Institut Jules Bordet, Anderlecht
  - Cliniques universitaires Saint-Luc, Brussels
  - UZ Gent, Ghent
  - Centre Hospitalier (CH) Jolimont, Haine-Saint-Paul
  - AZ Turnhout, Turnhout
- France (4):
  - Centre Hospitalier Universitaire (CHU) de Bordeaux, Bordeaux
  - Institut Paoli Calmettes, Marseille
  - Centre Hospitalier Universitaire (CHU) de Nice, Nice
  - Hôpital Saint-Louis, Paris
- Germany (5):
  - Universitätsklinikum Halle, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - University Hospital Jena, Jena
  - Universitätsklinikum Leipzig, Leipzig
  - Universitaetsklinikum Schleswig-Holstein, Lübeck
- Hungary (4):
  - Semmelweis Egyetem, Budapest
  - Del-Pesti Centrumkorhaz Orszagos Hematologiai es Infektologi, Budapest
  - szabolcs-szatmár-bereg megyei kórházak és egyetemi oktatókórház Jósa András Oktatókórház, Debrecen
  - Somogy Megyei KAposi Mor Oktato Korhaz, Kaposvár
- Israel (5):
  - Rambam Health Care Campus, Haifa
  - Hadassah Medical Center Ein Kerem, Jerusalem
  - The Chaim Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center, Tel Aviv
  - Assaf Harofeh Medical Center AHMC, Tel Aviv
- Italy (5):
  - Universitaria Maggiore della Carità Novara, Novara, Piedmont
  - A.O.O.R. Villa Sofia Cervello, Palermo, Sicily
  - AOU Policlinico S.Orsola-Malpighi, Bologna
  - AORMN Hospital Hematology and BMT Center, Pesaro
  - AOUS Le Scotte, Siena
- Uniwersyteckie Centrum Kliniczne, Gdansk, Poland
- South Korea (4):
  - Inje University Busan Paik Hospital, Busan
  - Seoul National University Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea-Seoul St. Mary's Hospital, Seoul
- Spain (9):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario de Gran Canaria Doctor Negrin, Las Palmas
  - MD Anderson Cancer Center, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario Virgen de la Victoria de Málaga, Málaga
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Clínico Universitario de Valencia, Valencia
- United Kingdom (4):
  - Birmingham Heartlands Hospital, Birmingham
  - University Hospital of Wales, Cardiff
  - The Royal Marsden Hospital, London
  - Oxford University Hospitals NHS Trust, Churchill Hospital, Oxford